CLINICAL TRIAL: NCT02749968
Title: Intercostal Liposomal Bupivacaine for the Management of Blunt Chest Wall Trauma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Goodman, instructor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Droege 2016
Record Dates: First submitted 2016-04-18; First posted 2016-04-25 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Blunt Chest Wall Trauma; Rib Fracture; Sternal Fracture
MeSH Terms: conditions — Rib Fractures | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liposomal bupivacaine (Active Comparator): 1 mL of liposomal bupivacaine injected with a 25-G needle just below each affected rib by the intercostal neurovascular bundle in a paraspinal position
  Interventions: Drug: Liposomal bupivacaine
- 0.9% sodium chloride (Placebo Comparator): 1 mL of 0.9% saline injected with a 25-G needle just below each affected rib by the intercostal neurovascular bundle in a paraspinal position
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: Liposomal bupivacaine — 1 mL of liposomal bupivacaine injected with a 25-G needle just below each affected rib by the intercostal neurovascular bundle in a paraspinal position
  Arms: Liposomal bupivacaine
Drug: 0.9% sodium chloride — 1 mL of 0.9% saline injected with a 25-G needle just below each affected rib by the intercostal neurovascular bundle in a paraspinal position
  Other Names: 0.9% saline
  Arms: 0.9% sodium chloride

SUMMARY:
This is a study of liposomal bupivacaine for pain control in patients with blunt chest wall trauma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of liposomal bupivacaine to provide analgesia via paravertebral intercostal nerve block following significant blunt chest trauma, minimizing adverse outcomes, length of stay and overall narcotic use. The primary outcome of the study is to compare requirements between the bupivacaine group and a standard-of-care group.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated length of stay of at least 72 hours
* Blunt chest wall trauma with two or more rib or sternal fractures
* Demonstrated ability to achieve > 50% predicted inspiratory capacity based on ideal body weight using IS within the first 24 hours of admission

Exclusion Criteria:

* Known allergy to bupivacaine
* Respiratory failure requiring intubation within 24 hours prior to enrollment
* Known or suspected atrioventricular nodal blockade process requiring cardiology evaluation or pacemaker placement
* Hemodynamic instability (defined as new intravenous vasopressor or inotrope requirement or mean arterial pressure < 55 mmHg)
* Signs of active myocardial ischemia or non-ST elevation MI
* > 20 rib fractures
* Weight < 50 kg or > 150 kg
* Pregnancy
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Goodman, MD, Principal Investigator — Department of Surgery, University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallen TE, Singer KE, Makley AT, Athota KP, Janowak CF, Hanseman D, Salvator A, Droege ME, Strilka R, Droege CA, Goodman MD. Intercostal liposomal bupivacaine injection for rib fractures: A prospective randomized controlled trial. J Trauma Acute Care Surg. 2022 Feb 1;92(2):266-276. doi: 10.1097/TA.0000000000003462. PMID 34789700

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: To achieve an 80% power with an alpha of 0.05, the goal enrollment was 200 patients. Interim analyses were performed after 50 patients further providing evidence to support the 200 patient goal for enrollment. Due to changes in analgesia protocols away from epidural catheters and a change in exclusion criteria to include those who were candidates for surgical stabilization of rib fractures, as well as the COVID-19 pandemic, enrollment was stopped at 100 patients
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | 0.9% Sodium Chloride
Started | 50 | 50
Interim Analysis (Interim safety and efficacy analysis was performed after 25 patients were recruited to each arm.) | 25 | 25
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | 0.9% Sodium Chloride | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (18) | 61 (18) | 60 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 25 | 28 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 50 | 100
  Unknown or Not Reported | 0 | 0 | 0
Incentive spirometry [Mean (Standard Deviation); unit: Liters/min] | 17.8 (8.1) | 17.6 (6.6) | 17.7 (7.39)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Requirement at 24 Hours Post-randomization
Description: Opioid requirement (in morphine equivalents) at 24 hours post-randomization
Time Frame: 24 hours following randomization.
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | 0.9% Sodium Chloride
Number analyzed (Participants) | 50 | 50
morphine milligram equivalents | 38 (959) | 202 (691)

2. Primary Outcome: Opioid Requirement at 48 Hours Post-randomization.
Description: Opioid requirement (in morphine equivalents) at 48 hours post-randomization
Time Frame: 48 hours following randomization.
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | 0.9% Sodium Chloride
Number analyzed (Participants) | 50 | 50
morphine milligram equivalents | 298 (1036) | 82 (129)

3. Primary Outcome: Opioid Requirement at 72 Hours Post-randomization
Description: Opioid requirement (in morphine equivalents) at 72 hours post-randomization
Time Frame: 72 hours following randomization.
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | 0.9% Sodium Chloride
Number analyzed (Participants) | 50 | 50
morphine milligram equivalents | 413 (1714) | 116 (199)

4. Primary Outcome: Opioid Requirement at 96 Hours Post-randomization
Description: Opioid requirement (in morphine equivalents) at 96 hours post-randomization
Time Frame: 96 hours following randomization.
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine | 0.9% Sodium Chloride
Number analyzed (Participants) | 50 | 50
morphine milligram equivalents | 637 (2012) | 39 (56)

5. Secondary Outcome: Development of Pneumonia
Description: Development of pneumonia defined as >100,000 colony forming units/milliliter bacteria on bronchoalveolar lavage or clinically with leukocytosis, pulmonary infiltrate and fever with 96 hours post-randomization.
Time Frame: 96 hours following randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | 0.9% Sodium Chloride
Number analyzed (Participants) | 50 | 50
Participants | 3 | 1

6. Secondary Outcome: Self-reported Pain at 96 Hours Post-randomization
Description: Self-reported pain will be measured using the verbal NRS, a 0-10 ordinal scale. Pain assessments will be reported at 96 hours after enrollment, as this is the reported duration of effect for liposomal bupivacaine. Higher scores (10) indicate more pain, lower scores (0) indicate lower pain.
Time Frame: At 96 hours post-randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | 0.9% Sodium Chloride
Number analyzed (Participants) | 50 | 50
score on a scale | 6.32 (2.73) | 6.44 (2.93)

ADVERSE EVENTS:
Time Frame: 96 hours
Arm/Group | Liposomal Bupivacaine | 0.9% Sodium Chloride
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 4/50 | 2/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liposomal Bupivacaine (N=50) | 0.9% Sodium Chloride (N=50)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
intubation (Respiratory, thoracic and mediastinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT02749968/Prot_SAP_000.pdf